CLINICAL TRIAL: NCT07098663
Title: A Phase 2a, Double-blind, Randomized, Placebo-controlled, Study to Assess Food Effect, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Oral Doses of MKP10241 in Healthy and Obese Adult Participants, With and Without Type 2 Diabetes Mellitus
Brief Title: Food Effect, Efficacy and Safety of MKP10241 in Healthy and Obese Adult Participants, With and Without Diabetes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mankind Pharma Limited (Industry)
Collaborators: Emerald Clinical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MKP10241-201
Record Dates: First submitted 2025-06-15; First posted 2025-08-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM); Food Effect; Safety and Tolerability; Obesity
Keywords: MKP10241; Safety and tolerability of MKP10241; Pharmacokinetics and Pharmacodynamics of MKP10241; Management of T2DM with MKP10241; Management of Obesity with MKP10241
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Intervention Model Description: Part 1 and Part 2 (Cohort 1) of the study will run in parallel. Part 3 will be a randomized, double-blind, placebo-controlled, Multiple ascending dose study.
Masking Description: Part 1 of the study is Open Label but Part 2 and 3 is a double blind ,in which participants/care providers/investigators/outcomes assessors, etc are blinded to study intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1- MKP10241 400 mg (Experimental): Participants will receive MKP10241 400 mg on Day 1 and Day 8.
  Interventions: Drug: MKP10241
- Part 1 - Placebo (Placebo Comparator): Participants will receive placebo 400 mg on Day 1 and Day 8.
  Interventions: Drug: Placebo
- Part 2 - MKP10241 200 mg, 300 mg and 400 mg (Experimental): Participants will receive MKP10241 200 mg, 300 mg and 400 mg daily from Day 1 to Day 28
  Interventions: Drug: MKP10241
- Part 2 - Placebo (Placebo Comparator): Participants will receive placebo daily from Day 1 to Day 28
  Interventions: Drug: Placebo
- Part 3 - MKP10241 300 mg and 400 mg (Experimental): Participants will receive MKP10241 300 mg and 400 mg daily from Day 1 to Day 28
  Interventions: Drug: MKP10241
- Part 3 - Placebo (Placebo Comparator): Participants will receive placebo daily from Day 1 to Day 28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MKP10241 — Oral liquid suspension of unit dose strength 6.6 mg/mL
  Arms: Part 1- MKP10241 400 mg; Part 2 - MKP10241 200 mg, 300 mg and 400 mg; Part 3 - MKP10241 300 mg and 400 mg
Drug: Placebo — Oral liquid suspension matched in appearance to MKP10241 at dosage strengths
  Arms: Part 1 - Placebo; Part 2 - Placebo; Part 3 - Placebo

SUMMARY:
The goal of this intervention study is to evaluate the safety, tolerability and pharmacokinetics (PK) and pharmacodynamics (PD) of multiple doses of MKP10241 in obese participants with and without T2DM in 3 parts. The main parameters it aims to answers are :

1. Does food effects the pharmacokinetic parameters following a single dose of MKP10241 in healthy participants?
2. Will multiple ascending doses of MKP10241 in obese participants with or without T2DM characterize changes in the plasma pharmacokinetic profile and pharmacodynamic effects?
3. What treatment emergent adverse events or discontinuation is experienced following single and multiple ascending doses of MKP10241 in healthy and obese participants with or without T2DM?

This study will be compared against a placebo which is matched in appearance to MKP10241 at dosage strengths.

Participants will:

1. Part 1: Take MKP10241 400 mg or Placebo on Day 1 and Day 8. Part 2: Take MKP10241 200 mg, 300 mg and 400 mg or Placebo daily from Day 1 to Day 28 Part 3: Take MKP10241 300 mg and 400 mg or Placebo daily from Day 1 to Day 28
2. Visit the clinical research unit for dose administration, admission or follow up.
3. Will be monitored by the Safety Monitoring Committee.

ELIGIBILITY:
Inclusion criteria

* Male or female participants between 18 to 60 years of age
* Considered healthy by the Investigator. Part 1: BMI of 18 to 30 kg/m2, and weight being not less than 50 kg. Part 2/3: BMI of ≥32 kg/m2
* Part 1/2: Fasting plasma glucose (FPG) between 3.9 mmol/L and 6.1 mmol/L. Part 3: FPG greater than or equal to 6.94 mmol/L and less than or equal to 14.43 mmol/L
* A nonsmoker/social smoker, defined as not having smoked more than 5 cigarettes or equivalent per day in the 3 months prior to Screening.
* Able to abstain from the consumption of alcohol and any alcohol-containing products from 48 hours before dosing to the End of Study Visit.
* Female participants must be of nonchildbearing potential or, if of childbearing potential, must agree to use 1 form of highly effective contraceptive method, plus an additional barrier method of contraception between signing consent
* Male participants who are sexually active must use a condom from Screening until at least 90 days after the last dose of study intervention (or be surgically sterile. Female partners of childbearing potential must use a highly effective method of contraception.
* Capable of giving signed Informed Consent
* Willing and able to adhere to study restrictions and to be confined at the CRU.
* Part 3: Participants with an established diagnosis of type 2 diabetes mellitus
* Part 3: Participants; type 2 diabetes mellitus must be managed by diet and exercise alone or by stable dose of metformin (for ≥2 months); the use of other antidiabetic therapies is prohibited

Exclusion criteria

* Clinically significant haematological findings at Screening.
* Hepatic impairment including aspartate aminotransferase (AST), alanine transaminase (ALT), or alkaline phosphatase ≥1.5 times upper limit of normal (ULN), total bilirubin ≥2.0 times ULN, albumin ≤3.0 g/L, serum amylase or lipase ≥1.5 times ULN at Screening.
* Renal impairment, such as creatinine ≥ULN, estimated glomerular filtration rate (eGFR) of ≤80 mL/minute/1.73m2 in adults, as calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* Positive polymerase chain reaction (PCR) test for severe-acute-respiratory-syndrome-related coronavirus (SARS-CoV-2)
* A history of non-febrile seizures.
* Positive pregnancy test result at Screening or on admission to the CRU,
* Any major surgery within 60 days prior to Screening, or planned major surgery during the study.
* Any history of malignant disease excluding surgically resected skin and in-situ cervical squamous cell or basal cell carcinoma.
* Suspected hypersensitivity to MKP10241 and any components of MKP10241 liquid suspension
* Any other condition which makes the participant unsuitable for study participation as judged by the Investigator or designee.
* Participant has any history or evidence of any clinically significant disease
* Prior or planned (during study period) bariatric surgery (e.g. gastric bands, gastroplasty Roux-e-Y gastric bypass) or ileal resection.
* Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, (DSM-V) substance use disorders and alcohol abuse within 12 months prior to Screening and/or positive alcohol breath test at Screening or admission.
* Positive result for drugs of abuse at Screening or admission.
* Use of live attenuated vaccines within 14 days prior to dosing
* The use of medications (other than paracetamol), including hormonal contraceptives
* Receipt of any other investigational medicinal product within one month or five half-lives (whichever is longer) prior to dosing.
* Clinically significant ECG findings: QTcF value ≥450 ms for males or ≥470 ms for females at Screening or Day -1
* Participants with a mean systolic blood pressure >140 mmHg, mean diastolic blood pressure >90 mmHg at Screening.
* Positive blood screen for human immunodeficiency virus antibody (HIV), hepatitis B surface antigen (HBsAg), syphilis, hepatitis C virus (HCV).
* Change in body weight of ≥ 10% within 3 months prior to the Screening visit.
* Donation or blood collection of more than 1 unit (approximate 450 mL) of blood (or blood products, plasma) or acute loss of blood during the 30 days prior to Screening.
* Part 3: Type 1 diabetes mellitus, maturity-onset diabetes of the young, or other forms of diabetes.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-04-17 (Estimated)

PRIMARY OUTCOMES:
Part 1 - Food effect of single dose of MKP10241 on Maximum concentration of drug (Cmax) | 18 days
  Maximum concentration (Cmax) following a single 400 mg dose of MKP10241 under fasting and fed condition
Part 1 - Food effect of single dose of MKP10241 on Apparent total clearance of drug (CL/F) | 18 days
  Total Clearance of the drug following a single 400 mg dose of MKP10241 under fasting and fed conditions
Part 1 - Food effect of single dose of MKP10241 on Time to maximum concentration (Tmax) | 18 days
  Time to maximum concentration (Tmax) following a single 400 mg dose of MKP10241 under fasting and fed condition
Part 1 - Food effect of single dose of MKP10241 on elimination half life (t1/2 ) | 18 days
  Elimination Half life (t1/2) following a single 400 mg dose of MKP10241 under fasting and fed conditions
Part 1 - Food effect of single dose of MKP10241 on lag time (Tlag) | 18 days
  Delay between the time of dosing and the time of appearance of the drug concentration in sampling (Tlag) for single 400 mg dose of MKP10241 under fasting and fed conditions
Part 1 - Food effect of single dose of MKP10241 on Apparent Volume of distribution of drug (V/F) | 18 days
  Apparent Volume of distribution of drug(V/F) following a single 400 mg dose of MKP10241 under fasting and conditions
Part 1 - Food effect of single dose of MKP10241 on Area under the curve from time 0 to 24hrs - AUC (0-24h) | 18 days
  Area under the plasma concentration time curve from time 0 to 24hrs - AUC(0-24h) following a single 400 mgMKP10241 under fasting and fed conditions
Part 1 - Food effect of single dose of MKP10241 on AUC(0-last) | 18 days
  Area under the curve from time 0 to the last value above the limit of quantification AUC(0-last) following a single dose of MKP10241 under fasting and fed conditions
Part 1 - Food effect of single dose of MKP10241 on AUC(0-inf) | 18 days
  Area under the curve from time 0 extrapolated to infinity AUC(0-inf) following a single 400 mg dose of MKP10241 fasting and fed conditions
Part 2 - To evaluate the incidence of treatment emergent adverse events and participant tolerance of MKP10241 following multiple doses in obese participants | 35 days
  It will be measured based on the Treatment emergent adverse events which includes significant changes in examination, blood and urine analysis, vital signs and ECG etc. Treatment discontinuation for any reason considered as intolerant.
Part 3 - To evaluate the incidence of treatment emergent adverse events and participant tolerance of MKP10241 following multiple doses in obese participants with T2DM. | 35 days
  It will be measured based on the Treatment emergent adverse events which includes significant changes in examination, blood and urine analysis, vital signs and ECG etc. Treatment discontinuation for any reason considered as intolerant.

SECONDARY OUTCOMES:
Part 1 - To evaluate the incidence of treatment emergent adverse events and of MKP10241 following a single dose administered orally under fasting and fed conditions. | 18 days
  It will be measured based on the Treatment emergent adverse events which includes significant changes in examination, blood and urine analysis, vital signs and ECG etc.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants the below will be measured:
  Change in Heart Rate in beats per minute
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in the below will be measured:
  Change in body weight in kilograms
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in the below will be measured:
  Change in BMI in kilograms per meter square
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants. | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in the below will be measured:
  Change in mid-abdominal circumference in centimeters
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Baseline to Day 28
  Pharmacodynamic parameters - Heart rate in beats per minute
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in the below will be measured:
  Change in body weight in kilograms
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in the below will be measured:
  • Change in Body Mass index in kilogram per meter square
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants given in below will be measured:
  Change in mid-abdominal circumference in centimeters
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Baseline to Day 28
  Pharmacodynamic parameters - To evaluate surrogate markers of efficacy and mechanism of action in obese participants the below will be measured:
  Change in Blood Pressure in millimeters of mercury (mmHg)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | From screening visit to day 29
  Pharmacodynamic parameters: Oral Glucose Tolerance Test
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 7, 14, 21 and 28
  Pharmacodynamic parameters - Fasting plasma glucose pre-dose on Days 1, 7, 14, 21 and 28.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters -
  Total insulin levels pre-dose, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4 hours, 6.0 hours, 8.0 hours, and Day 1, 28 and 24 hours post-dose on Day 2 and 29.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants with T2DM. | Day 1, 2 , 28 and 29
  Pharmacodynamic parameters -
  GLP-1 (active and total) levels pre-dose, 0.25 hours, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, and 12 hours on Day 1, 28 and 24 hours post-dose on Day 2 and 29.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants with T2DM. | At Baseline,Day 1, 7, 14, 21 and Day 28
  Pharmacodynamic parameters - Total cholesterol levels
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants. | At baseline and Day 28
  Pharmacodynamic parameters - Lipase
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | At baseline and Day 28
  Pharmacodynamic parameters - Total amylin
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | At baseline and Day 28
  Pharmacodynamic parameters - C-Reactive Protein
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | At baseline and Day 28
  Pharmacodynamic parameters - Hepatic transaminases
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Baseline to Day 28
  Pharmacodynamic parameters - Blood Pressure
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 7, 14, 21 and 28.
  Pharmacodynamic parameters - Fasting plasma glucose pre-dose on Days 1, 7, 14, 21 and 28.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1,2,28 and 29
  Pharmacodynamic parameters - Total Insulin pre-dose, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - Glucagon levels pre-dose, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hour, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - GLP 1 pre-dose, 0.25 hours, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - C peptide pre-dose, 0.25 hours, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0hours, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - Total Glucose-dependent Insulinotropic Polypeptide pre-dose, 0.25 hours, 0.5 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - total amount of Peptide YY (PYY) pre-dose, 0.25 hours, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - Leptin pre-dose, 0.25 hours, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | At Baseline,Day 1, 7, 14, 21 and Day 28
  Pharmacodynamic parameters - Total cholesterol levels
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | At baseline and Day 28
  Pharmacodynamic parameters - total amylin
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM | At baseline and Day 28
  Pharmacodynamic parameters - C-Reactive Protein
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | At baseline and Day 28
  Pharmacodynamic parameters - Hepatic transaminases
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Maximum concentration (Cmax)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Total Clearance of the drug
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Time to maximum concentration(Tmax)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation -Elimination Half life (t1/2)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Delay between the time of dosing and the time of appearance of the concentration in sampling (Tlag)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Apparent Volume of distribution of drug(V/F)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Area under the plasma concentration time curve from time 0 to 24hr
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Area under the curve from time 0 to the last value above the limit of quantification AUC(0-last)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | 35 days
  Pharmacokinetic parameter evaluation - Area under the curve from time 0 extrapolated to infinity AUC(0-inf)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Maximum concentration (Cmax)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Total Clearance of the drug
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Time to maximum concentration(Tmax)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Elimination Half life (t1/2)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Delay between the time of dosing and the time of appearance of the concentration in sampling (Tlag)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Apparent Volume of distribution of drug(V/F)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Area under the plasma concentration time curve from time 0 to 24hours
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | 35 days
  Pharmacokinetic parameter evaluation - Area under the curve from time 0 to the last value above the limit of quantification AUC(0-last)
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM | 35 days
  Pharmacokinetic parameter evaluation - Area under the curve from time 0 extrapolated to infinity AUC(0-inf)
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 2, 28 and 29
  Pharmacodynamic parameter - Glucagon levels pre-dose, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours and 12 hours on Day 1 and 28 and 24 hours post-dose on Day 2 and 29
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - C-peptide levels pre-dose, 0.25 hours, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hour, 4.0 hour, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 2,28 and 29
  Pharmacodynamic parameters - total GIP levels pre-dose, 0.25 hours, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hours, 4.0 hour, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - total PYY levels pre-dose, 0.25 hours, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hour, 4.0 hour, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - leptin levels pre-dose, 0.25 hours, 0.5 hours, 1.0 hour, 2.0 hours, 3.0 hours, 4.0 hour, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29.
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | Day 1, 2, 28 and 29
  Pharmacodynamic parameters - glycated hemoglobin HbA1c pre-dose, 0.25 hours, 0.5 hours, 1.0 hours, 2.0 hours, 3.0 hours, 4.0 hours, 6.0 hours, 8.0 hours, and 12 hours on Day 1 and 28, and 24 hours post-dose on Day 2 and 29
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | At baseline and Day 28
  Pharmacodynamic parameters - Lipase
Part 2 - Pharmacokinetics and Pharmacodynamics of MKP10241 following multiple doses in obese adult participants with T2DM. | At Baseline,Day 1, 7, 14, 21 and Day 28
  Pharmacodynamic parameters - Triglyceride
Part 3 - Pharmacokinetic and Pharmacodynamic effects of MKP10241 following multiple doses administration in obese adult participants with T2DM. | At Baseline,Day 1, 7, 14, 21 and Day 28
  Pharmacodynamic parameters - Triglyceride

OTHER OUTCOMES:
Part 2 - Impact of multiple doses of MKP10241 administered to obese participants without T2DM on participant Hunger and Satiety Visual Analogue Scale | Day 14 and Day 28 from baseline
  Will be checked for change in participant Hunger and Satiety VAS score on Day 14 and Day 28 from baseline Participants will be asked to make a mark on a scale to indicate their hunger levels. The distance along line where the participant made their mark will be used as the measure.
  The distance in mm the participant marks on the scale will be used as a quantitative measure.Shorter means not hungry at all and higher means more hungry.
Part 2 - Impact of multiple doses of MKP10241 administered to obese participants without T2DM on participant Visceral fat | Baseline to Day 32
  Visceral fats will be measured by MRI-PDFF. The change in magnetic resonance derived proton density visceral fat fraction i.e. percentage of fat in the whole abdominal region will be measured.
Part 3 - Impact of multiple doses of MKP10241 administered to obese participants with T2DM on participant Hunger levels and Satiety Visual Analogue Scale. | Day 14 and Day 28 from baseline.
  Will be checked for change in participant Hunger and Satiety VAS score on Day 14 and Day 28 from baseline(Day- 1) Participants will be asked to make a mark on a scale to indicate their hunger levels. The distance along line where the participant made their mark will be used as the measure. The distance in mm the participant marks on the scale will be used as a quantitative measure.
  Shorter means not hungry at all and higher means more hungry.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hall, MBBS, FRACP, Principal Investigator — Veritus Research
Locations (1):
- Veritus Research, Bayswater, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No